CLINICAL TRIAL: NCT05420402
Title: Effect of Different Administrations of Propofol on Emergence Agitation in Preschool Children Undergoing Ambulatory Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiaxiang Chen (Other)
Responsible Party: Sponsor-Investigator, Jiaxiang Chen, Principal Investigator, Shantou University Medical College
Organization: Shantou University Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SZanes0712
Record Dates: First submitted 2022-06-01; First posted 2022-06-15 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-10

CONDITIONS: Anesthesia; Surgery
Keywords: Emergence Agitation; Ambulatory Surgery; Preschool Children; Propofol
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bolus group A (Active Comparator): 42 participants will receive 1 mg/kg intravenous bolus of propofol 3 min before the end of surgery.
  Interventions: Drug: Propofol bolus
- Continuous infusion group (Active Comparator): 42 participants will receive 1 mg/kg continuous intravenous pumping of propofol 3 minutes before the end of the operation, and the pumping time was 3 minutes.
  Interventions: Drug: Propofol continuous infusion
- Bolus group B (Active Comparator): 42 participants will receive 1 mg/kg intravenous bolus of propofol at the end of surgery.
  Interventions: Drug: Propofol bolus
- Blank Comparator group (No Intervention): 42 participants will not receive propofol

INTERVENTIONS:
Drug: Propofol bolus — A bolus dose of propofol 1 mg/kg was administered intravenously at 3 minutes before the end of the surgery.
  Other Names: 3 minutes before the end of the surgery
  Arms: Bolus group A
Drug: Propofol continuous infusion — 1 mg/kg propofol was started by continuous infusion 3 minutes before the end of surgery, and the infusion time was 3 minutes.
  Other Names: 3 min intravenous pumping
  Arms: Continuous infusion group
Drug: Propofol bolus — A bolus dose of propofol 1 mg/kg was administered intravenously at the end of the surgery.
  Other Names: at the end of the surgery
  Arms: Bolus group B

SUMMARY:
This study evaluates the influence of different dose and methods of propofol on emergence agitation(EA) through a randomized controlled trial when preschool children undergoing ambulatory surgery of inguinal hernia.

DETAILED DESCRIPTION:
Emergency agitation (EA) is the manifestation of excitement, high irritability, intense struggle, and increased blood pressure and heart rate during the recovery period of general anesthesia. It is a common adverse reaction after general anesthesia. The incidence in preschool children is 10%-80%, which is currently considered to be mainly related to factors such as the use of inhalation anesthetics, pain stimulation, drug types, surgical methods, and environmental changes. EA not only increases children's risks, such as drains and dehiscence, but also increases caregiver stress and reduces parental satisfaction with the method of anesthesia.

This trial is a randomized single-blind clinical trial. The padiatric patients were randomly divided into 4 groups.The block randomization is generated by statistical professionals using SAS9.2 software. The block size is fixed at 8 and randomly changed. Each random number and the corresponding assignment result are placed in a sealed in a transparent envelope. The investigator is responsible for including subjects according to the requirements of the program. When the subjects meet the inclusion criteria but not the exclusion criteria, the field staff will open the envelopes in order to group them.The clinical anesthesia and data statistical analysis were completed by different anesthesiologists and participants.

The four groups of children were fasted for 6 hours and 2 hours before operation, and no preoperative medication was given. After the children were awake and entered the room, the heart rate (HR), non-invasive blood pressure (NIBP), pulse oxygen saturation (SpO2), respiratory rate (RR) and end-tidal carbon dioxide partial pressure (PetCO2) were continuously monitored. Both groups were given routine standard anesthesia induction: intravenous injection of midazolam at 0.05-0.1 mg/kg of predicted body weight (PBW), propofol at 2-4 mg/kg of PBW, and remifentanil at 1-2 ug/kg of PBW, rocuronium at 0.5-1mg/kg of PBW.After adequate pre-oxygenation,laryngeal mask was placed.Anesthesia was maintained by inhalation of 2%-3% sevoflurane and continuous pumping of remifentanil at 0.2-0.4ug/kg/min remifentanil, with an oxygen flow of 2L/min. The tidal volume method was used in all mechanical ventilation. The tidal volume was between 6 and 8 mL/kg, the respiratory rate was between 18 and 24 breaths/min, and the PetCO2 was maintained between 30 and 35 mmHg. Three minutes before the end of surgery, the oxygen flow was adjusted to 6 L/min, sevoflurane was stopped, and the infusion of remifentanil was stopped. At the end of the operation, the children in all groups received local infiltration anesthesia with 0.3% ropivacaine around the incision by the surgeon.

The children in group A were given 1 mg/kg propofol intravenous bolus 3 minutes before the end of the operation.Children in group B were given continuous pumping of 1 mg/kg propofol 3 minutes before the end of the operation, and the infusion time was 3 minutes. Children in group C 1 mg/kg propofol was given intravenously at the end of the operation. Children in group D were not given propofol and served as a blank control group.

All data were collected, aggregated and maintained by a single investigator.The primary outcome measure was the anesthesia emergence delirium scale (PAED). The observation was performed during the recovery period of the child, and the child opened his eyes voluntarily to the stage of complete recovery of consciousness. Mainly from the three aspects of eye contact, behavior and consciousness, the total score is 20 points. 15 points for severe agitation.In addition, the indicators we collected also include age, gender, weight, ASA classification, operation method, operation time, discharge time and occurrence of adverse reactions and so on.

The full analysis set was used for analysis. According to the basic principle of Intention-to-Treat (ITT), the analysis of the main indicators includes all randomized subjects, regardless of whether they completed the trial or not, that is, subjects who were lost to follow-up should also be included in the statistical analysis. Statistical software SPSS 26.0 was used for data processing and statistical analysis. Shapiro-Wilk test was first performed on the data, and continuous variable data (such as blood pressure, heart rate, driving pressure, oxygenation index, etc.) were determined to use Analysis of variance or Kruskal-Wallis H test according to their normal distribution. Categorical variables (such as age,incidence of EA, etc.) were tested by χ² test, Fisher's exact test, and the results were expressed as mean ± standard deviation (SD), percentage (%) or median (interquartile range, IQR), P <0.05 is statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-5 years
* ASA classification 1
* Written informed consent
* Children undergoing ambulatory surgery of inguinal hernia
* The operation will take no more than 20 minutes

Exclusion Criteria:

* Allergic to drugs used in the study
* Neurological disorders
* Congenital heart insufficiency
* Recent respiratory illness

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of emergence agitation | Within up to 30 minutes after operation
  Pediatric anesthesia emergence delirium scale (PAED). The total score is 20 points.A score of 10 or above is considered as EA and 15 or above is considered as severe EA.

SECONDARY OUTCOMES:
length of hospital stay | 1 day post surgery
  The length of time the patient took from leaving the operating room to being discharged from the hospital.
The occurrence of adverse reactions | Within up to 30 minutes after operation
  These include both gastrointestinal and respiratory reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Children's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication and with no end date
Access Criteria: Researchers who provide a methodologically sound proposal To achieve aims in the approved proposal.
  Proposals should be directed to Dr Jiaxiang Chen; e-mail address:cjxanes@163.com
  To gain access, data requestors will need to sign a data Access agreement.

REFERENCES:
- [Result] Fabricant PD, Seeley MA, Rozell JC, Fieldston E, Flynn JM, Wells LM, Ganley TJ. Cost Savings From Utilization of an Ambulatory Surgery Center for Orthopaedic Day Surgery. J Am Acad Orthop Surg. 2016 Dec;24(12):865-871. doi: 10.5435/JAAOS-D-15-00751. PMID 27792057
- [Result] Shinnick JK, Short HL, Heiss KF, Santore MT, Blakely ML, Raval MV. Enhancing recovery in pediatric surgery: a review of the literature. J Surg Res. 2016 May 1;202(1):165-76. doi: 10.1016/j.jss.2015.12.051. Epub 2016 Jan 12. PMID 27083963
- [Result] Moore AD, Anghelescu DL. Emergence Delirium in Pediatric Anesthesia. Paediatr Drugs. 2017 Feb;19(1):11-20. doi: 10.1007/s40272-016-0201-5. PMID 27798810
- [Result] Kanaya A. Emergence agitation in children: risk factors, prevention, and treatment. J Anesth. 2016 Apr;30(2):261-7. doi: 10.1007/s00540-015-2098-5. Epub 2015 Nov 24. PMID 26601849
- [Result] Jacob Z, Li H, Makaryus R, Zhang S, Reinsel R, Lee H, Feng T, Rothman DL, Benveniste H. Metabolomic profiling of children's brains undergoing general anesthesia with sevoflurane and propofol. Anesthesiology. 2012 Nov;117(5):1062-71. doi: 10.1097/ALN.0b013e31826be417. PMID 22929729
- [Result] Chidambaran V, Costandi A, D'Mello A. Propofol: a review of its role in pediatric anesthesia and sedation. CNS Drugs. 2015 Jul;29(7):543-63. doi: 10.1007/s40263-015-0259-6. PMID 26290263
- [Result] Wu X, Cao J, Shan C, Peng B, Zhang R, Cao J, Zhang F. Efficacy and safety of propofol in preventing emergence agitation after sevoflurane anesthesia for children. Exp Ther Med. 2019 Apr;17(4):3136-3140. doi: 10.3892/etm.2019.7289. Epub 2019 Feb 20. PMID 30930979
- [Result] van Hoff SL, O'Neill ES, Cohen LC, Collins BA. Does a prophylactic dose of propofol reduce emergence agitation in children receiving anesthesia? A systematic review and meta-analysis. Paediatr Anaesth. 2015 Jul;25(7):668-76. doi: 10.1111/pan.12669. Epub 2015 Apr 27. PMID 25917689
- [Result] Malarbi S, Stargatt R, Howard K, Davidson A. Characterizing the behavior of children emerging with delirium from general anesthesia. Paediatr Anaesth. 2011 Sep;21(9):942-50. doi: 10.1111/j.1460-9592.2011.03646.x. Epub 2011 Jul 5. PMID 21726352
- [Result] Bajwa SA, Costi D, Cyna AM. A comparison of emergence delirium scales following general anesthesia in children. Paediatr Anaesth. 2010 Aug;20(8):704-11. doi: 10.1111/j.1460-9592.2010.03328.x. PMID 20497353
- [Derived] Chen J, Shi X, Hu W, Lin R, Meng L, Liang C, Ma X, Xu L. Comparing different administration methods of subanaesthetic propofol to mitigate emergence agitation in preschool children undergoing day surgery: a double-blind, randomised controlled study. BMJ Paediatr Open. 2025 Mar 15;9(1):e002376. doi: 10.1136/bmjpo-2023-002376. PMID 40090678